CLINICAL TRIAL: NCT04034628
Title: Improving the Outcomes of Peritoneal Dialysis (PD) Catheter Insertion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Matthew Oliver, Associate Professor, Sunnybrook Health Sciences Centre
Other Study IDs: 160-2019
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Peritoneal Dialysis Access Failure; Peritoneal Dialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic insertion: Individuals who undergo laparoscopic PD catheter insertion
  Interventions: Device: Peritoneal Catheter Insertion - Laparoscopic; Device: Peritoneal Catheter Insertion - Percutaneous
- Percutaneous insertion: Individuals who undergo percutaneous PD catheter insertion by either a nephrologist or radiologist.
  Interventions: Device: Peritoneal Catheter Insertion - Laparoscopic; Device: Peritoneal Catheter Insertion - Percutaneous

INTERVENTIONS:
Device: Peritoneal Catheter Insertion - Laparoscopic — Insertion of a Peritoneal Catheter into the abdomen for the purposes of treating kidney failure
Device: Peritoneal Catheter Insertion - Percutaneous — Insertion of a Peritoneal Catheter into the abdomen for the purposes of treating kidney failure

SUMMARY:
Peritoneal dialysis (PD) is actively promoted as the preferred form of dialysis for patients with kidney failure. However, 1 in 5 patients will experience a signification catheter insertion-related PD catheter complication in the first 6 months following insertion. Little is known about the patient-, operator-, and center-level factors that influence PD catheter complications. There is a need to identify key modifiable practices to focus randomized trials and quality improvement efforts. We will leverage prior funding, a custom-built data collection platform, pilot data, and a group of engaged stakeholders, partners, and knowledge users to: a) Determine if method of insertion is associated with PD catheter complications b) Identify operator/center characteristics and practices associated with PD catheter complications c) Use a data-driven approach to achieve expert consensus on optimal practices for PD catheter insertion and care.

DETAILED DESCRIPTION:
Patient population and setting. We will identify all patients undergoing their first PD catheter insertion during the study period, at 20 participating centers in Canada and the USA (see Appendix 1). A total of 800 cases have been captured to date during our pilot study and an additional 1,520 cases will be accrued over a 30-month period, for a total sample size of 2,320 PD catheter insertions. We will attempt to collect information about consecutive patients undergoing PD catheter attempts/insertions in order to accurately measure local performance. However if a waiver of consent cannot be obtained at participating centers, then non-consecutive patients will be enrolled.

Inclusion criteria: patients must be 18 years of age or older; have advanced chronic kidney disease; have chosen PD as their intended treatment modality; and undergone their first PD catheter placement during the study period.

Exclusion criteria: patients who intend to transfer to another PD program or who are scheduled to receive a transplant within 3 months of the start of PD therapy will be excluded. Data source: ISPD Catheter Registry. The ISPD Catheter Registry is a web-based data collection tool that was custom-built for this project. It was developed based on a patented approach (Canadian patent #2,666,569; issued 2/28/2017)

Patient-level variables for our models will include baseline demographic (age, sex), comorbidity [body mass index (BMI), chronic kidney disease (dialysis-dependent vs. not), diabetes mellitus, cardiovascular disease (coronary artery disease, peripheral vascular disease, cerebrovascular disease), congestive heart failure, respiratory disease, liver disease, abdominal scarring, history of abdominal hernias], laboratory (hemoglobin, albumin), and medication variables (use of anticoagulants, antiplatelet, immunosuppressive medications).

Operator variables include operator volume, advanced training in PD catheter insertion and years of experience placing PD catheters.

Primary outcome: PD catheter complications. Our primary outcome will be the composite of the need for interventional procedures, emergency room visits and hospitalizations, reduction in time on PD, or discontinuation of PD therapy due to insertion-related PD catheter complications.

Sample size of 2,000 patients will provide 80% power to detect a 25% relative reduction in the risk of our primary outcome in those undergoing laparoscopic insertion of their catheter, across a range of possible ICC values. In order to guard against a larger than anticipated intra-class correlation coefficient(up to 0.001), we will target a sample size of 2,320 patients

ELIGIBILITY:
Inclusion Criteria:patients must be 18 years of age or older; have advanced chronic kidney disease; have chosen PD as their intended treatment modality; and undergone their first PD catheter placement during the study period.

Exclusion Criteria:patients who intend to transfer to another PD program or who are scheduled to receive a transplant within 3 months of the start of PD therapy will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will identify all patients undergoing their first PD catheter insertion during the study period, at 20 participating centers in Canada and the USA (see Appendix 1).
  A total of 800 cases have been captured to date during our pilot study and an additional 1,520 cases will be accrued over a 30-month period, for a total sample size of 2,320 PD catheter insertions. We will attempt to collect information about consecutive patients undergoing PD catheter attempts/insertions in order to accurately measure local performance. However if a waiver of consent cannot be obtained at participating centers, then non-consecutive patients will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 2320 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Insertion related complications | 1 year following the start of PD therapy
  Complications (exit site leak, flow restriction, pain, infection, bleeding) likely associated with the method of insertion

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Oliver, MD MHS, Principal Investigator — University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We would be willing to collaborate depending on the project.